CLINICAL TRIAL: NCT00168649
Title: The Effect of Vitamin A on the Response to Endotoxin
Brief Title: Vitamin A and Response to Endotoxin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bandim Health Project (Other)
Collaborators: Uppsala University Hospital (Other); Institute for Human Nutrition, Royal Veterinary School, Copenhagen, Denmark (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: 9583-2625-VITA-LPS; 9583-2625
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2013-11-15 (Estimated); Status verified 2013-11

CONDITIONS: TNF-alfa; Endotoxin Levels
Keywords: Vitamin A; Endotoxin; TNF-alfa
MeSH Terms: interventions — Vitamin A

INTERVENTIONS:
Drug: Vitamin A

SUMMARY:
Vitamin A given as treatment and pre-treatment has reduced the severity of symptoms after infusion with endotoxin in several animal models. We intend to examine the effect of vitamin A as pre-treatment on the response to endotoxin in humans. We furthermore wish to examine the long-term effects of vitamin A on the response to endotoxin. We hypothesise that vitamin A decreases endotoxin levels and TNF-alfa responses.

DETAILED DESCRIPTION:
Vitamin A given as treatment and pre-treatment has reduced the severity of symptoms after infusion with endotoxin in several animal models. We intend to examine the effect of vitamin A as pre-treatment on the response to endotoxin in humans. As studies in children in low-income countries have indicated that vitamin A has long-term effects on the immune system, we furthermore wish to examine the long-term effects of vitamin A on the response to endotoxin. This will be done in an established model using infusion with endotoxin to male human volunteers. We hypothesise that vitamin A decreases endotoxin levels and TNF-alfa responses. Furthermore, we hypothesise that it reduces oxidative stress and injury.

ELIGIBILITY:
Inclusion Criteria: Healthy, male, between 18 and 35 years of age, non-smoker, no medicine, no infections in preceding 14 days

Exclusion Criteria:

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40
Dates: Start 2005-06; Study Completion 2014-06

PRIMARY OUTCOMES:
Endotoxin levels
TNF-alfa levels

SECONDARY OUTCOMES:
Measures of oxidative injury and stress
Retinol and beta-caroten levels
Haematological values
Clinical markers

CONTACTS AND LOCATIONS:
Overall Officials: Bente K Pedersen, MD, DMSc, Study Director — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Department M7641, Copenhagen, Denmark